CLINICAL TRIAL: NCT00539994
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Efficacy of Retapamulin Ointment, 1% Applied Twice Daily for 3 or 5 Days to the Anterior Nares of Healthy Adult Subjects Nasally Colonized With Staphylococcus Aureus
Brief Title: Retapamulin Ointment in Healthy Adults Nasally Colonized With Staphylococcus Aureus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ALB110247
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Results first posted 2010-08-20 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-11

CONDITIONS: Infections, Bacterial
Keywords: Altabax; SB-275833; retapamulin; nasal colonization; PK; tolerability; safety; efficacy
MeSH Terms: conditions — Bacterial Infections | interventions — retapamulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment B (Experimental): 200mg BID retapamulin 5 days
  Interventions: Drug: Retapamulin
- Treatment C (Placebo Comparator): 200mg BID placebo 5 days
  Interventions: Drug: Placebo
- Treatment A (Experimental): 200mg BID retapamulin 3 days and placebo BID 2 days for a total of 5 days
  Interventions: Drug: retapamulin

INTERVENTIONS:
Drug: retapamulin — 200mg BID retapamulin 3 days
  Arms: Treatment A
Drug: Retapamulin — 200mg BID retapamulin 5 days
  Arms: Treatment B
Drug: Placebo — 200mg BID placebo 5 days
  Arms: Treatment C

SUMMARY:
This is a Phase I/IIa randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK, and efficacy of Retapamulin ointment, 1% applied twice daily for 3 or 5 days to the anterior nares of healthy adult subjects who are nasally colonized with S. aureus. Approximately 57 healthy subjects who are nasal carriers of S. aureus will be enrolled and stratified in a 2:1 ratio so that at least 38 persistent carriers and 19 intermittent carriers complete the study. Each eligible subject will participate in three screening visits, a treatment period, and two follow-up visits. Each subject's participation in the study will be approximately 6 to 10 weeks from screening to the last follow-up visit. Subjects will participate in up to three screening visits to determine S. aureus culture positivity and colonization status.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 and 65, inclusive. A female is eligible to enter and participate in this study if she is non-pregnant, nonlactating and if she is of:

  * non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy or documented tubal ligation or post-menopausal females defined as being amenorrheic for greater than one year and having follicle stimulating hormone (FSH) levels consistent with menopause.
  * child-bearing potential has a negative pregnancy test at screening. In addition, she must be willing to abstain from sexual intercourse or must use a nonhormone contraception such as an IUD or diaphragm with spermicide, in addition to having their male partner use condom/spermicide. This criterion must be followed from at least the commencement of her last normal period prior to the first dose of study medication or from screening (whichever is earlier) until completion of all follow-up procedures (33 days after the last dose of study medication).
* Body weight ≥ 50 kg for men and ≥ 45 kg for women and a body mass index (BMI) between 18.5 - 33 kg/m2.
* The subject is able to understand and comply with requirements, instructions and restrictions listed in the consent form.
* Signed and dated written informed consent prior to admission to the study.

Exclusion Criteria:

* Negative nasal culture for S. aureus on the first screen visit.
* Negative nasal cultures for S. aureus on second and third screen visits.
* Concurrent treatment with antimicrobials for an infection.
* MRSA decolonization attempt in the previous 6 months (prior treatment for a MRSA infection is not an exclusion criterion).
* Inability to take medications nasally.
* Nasal surgery in the previous 3 months.
* Evidence of active rhinitis, sinusitis, or upper respiratory infection.
* Within the judgment of the Principal Investigator and the Sponsor Medical Monitor, any clinically significant hematologic, endocrine, cardiovascular, hepatic, renal, gastrointestinal, and/or pulmonary disorder; any predisposing condition that might interfere with the absorption, distribution, metabolism, and/or excretion of drugs; or any clinically relevant abnormality identified on physical examination, 12-lead ECG, or clinical laboratories at screening. A single repeat for clinical laboratories or 12- lead ECG will be allowed to determine eligibility.
* The subject's systolic BP is outside the range of 90-150mmHg, or diastolic BP is outside the range of 45-95mmHg or HR is outside the range of 50-100 bpm for female subjects or 40-100 bpm for male subjects.
* Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* The use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety. Use of nasal medications is strictly prohibited from 7 days prior to the first screening visit and then 7 days prior to the 2nd screening visit through the final follow-up visit.
* Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
* The subject has a history of alcohol or substance abuse or dependence within 12 months of the study: History of regular alcohol consumption averaging > 7 drinks/wk for women or > 14 drinks/wk for men. 1 drink is equivalent to 12g alcohol = 5 oz (150ml) of wine or 12oz (360ml) of beer or 1.5 oz (45ml) of 80 proof distilled spirits within six months of screening.
* Positive for Human Immunodeficiency Virus (HIV) antibody, hepatitis B virus surface antigen or hepatitis C virus antibody at screening.
* Donation of blood in excess of 500 mL within 56 days prior to dosing. Note: This does not include plasma donation.
* The subject has a positive urine drug or alcohol screen.
* The subject has a history of illicit drug abuse or is unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Naderer OJ, Anderson M, Roberts K, Lou Y, Zhu J, Min S, Scangarella N, Shawar, R. Nasal Decolonization of Persistent Staphylococcus aureus Carriers with Twice Daily Retapamulin Treatment for 3 or 5 Days. Presentation Number L-1492. 48th ICAAC/46th IDSA Annual Meeting, Washington, DC, October 25-28, 2008.
- [Background] Naderer OJ, Anderson M, Roberts K, Scangarella N, Shawar R, Mundy LM. Case detection of Staphylococcus aureus colonization: screening of the anterior nares (AN) and throat (T). Presentation Number K-3353. 48th Interscience Conference on Antimicrobial Agents and Chemotheraty (ICAAC)/46th Infectious Diseases Society of America (IDSA) Annual Meeting, Washington, DC, October 25-28, 2008.
- [Background] Scangarella N, Naderer OJ, Anderson M, Roberts K, Sahm D, Shawar R. Antibacterial Activity of Retapamulin and Comparators Against Nasal and Pharyngeal Staphylococcus aureus Isolates Recovered from a Clinical Trial Investigating the Efficacy of Retapamulin in Nasal Decolonization. Presentation Number C1-3840. 48th ICAAC/46th IDSA Annual Meeting, Washington, DC, October 25-28, 2008.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: ALB110247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ALB110247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ALB110247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ALB110247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ALB110247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ALB110247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ALB110247 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Retapamulin 3 Days: Retapamulin ointment, 1% 200 mg BID 3 days and 200 mg Placebo BID for 2 days
- Retapamulin 5 Days: Retapamulin ointment, 1% 200 mg BID 5 days
- Placebo: Placebo 200 mg BID for 5 days
Period: Overall Study
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days | Placebo
Started | 23 | 19 | 15
Completed | 20 | 18 | 13
Not Completed | 3 | 1 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days | Placebo | Total
Number analyzed (Participants) | 23 | 19 | 15 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.8 (10.80) | 35.8 (11.16) | 33.7 (12.67) | 33.6 (11.36)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 6 | 2 | 14
  Male | 17 | 13 | 13 | 43
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 4 | 7 | 3 | 14
  Asian - East Asian Heritage | 0 | 0 | 1 | 1
  Asian - Japanese Heritage | 0 | 2 | 0 | 2
  Asian - South East Asian Heritage | 0 | 1 | 0 | 1
  White | 18 | 7 | 9 | 34
  Mixed Race | 1 | 2 | 2 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 22 | 18 | 13 | 53
Efficacy population by carrier type (persistent vs intermittent) [Number; unit: participants]
  Persistent, Intent-to-Treat | 17 | 16 | 13 | 46
  Intermittent, Intent-to-Treat | 1 | 2 | 0 | 3
  Excluded from analysis | 5 | 1 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Plasma Retapumulin Pharmacokinetic Parameters by Treatment at Days 1 and 3 Evaluated by Plasma AUC After Dosing
Description: Area under the plasma concentration curve (AUC) is used to calculate drug clearance and bioavailability using plasma concentration and time curve.
Time Frame: Days 1 and 3
Population: Pharmacokinetic (PK) Concentration Population - included all subjects who underwent plasma PK sampling
Measure: Mean (Standard Deviation); unit: ng.h /mL
Groups:
- Retapamulin 3 Days: Retapamulin ointment, 1% 200 mg BID 3 days and Placebo 2 days
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days
Number analyzed (Participants) | 14 | 10
ng.h /mL
  Day 1, n=5 and 2 | 0.8663 (1.77269) | 0.3816 (0.89226)
  Day 3, n=14 and 10 | 4.2802 (5.37822) | 2.0881 (3.47126)

2. Primary Outcome: Plasma Retapumulin Pharmacokinetic Parameters by Treatment at Day 5 Evaluated by Plasma AUC After Dosing
Description: as for outcome 1
Time Frame: Day 5
Population: Pharmacokinetic Concentration Population - included all subjects who underwent plasma PK sampling
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days
Number analyzed (Participants) | 0 | 9
ng.h/mL |  | 1.8883 (3.05391)

3. Primary Outcome: Plasma Retapumulin Pharmacokinetic Parameters by Treatment at Days 1 and 3 Evaluated by Plasma Cmax After Dosing
Description: Cmax is the peak serum concentration. Low value was not calculable, and High value was 2.74 ng/mL.
Time Frame: Days 1 and 3
Population: Pharmacokinetic Concentration Population - included all subjects who underwent plasma PK sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days
Number analyzed (Participants) | 16 | 10
ng/mL
  Day 1, n=10 and 3 | 0.4703 (0.34262) | 0.3538 (0.27237)
  Day 3, n=16 and 10 | 0.7893 (0.56984) | 0.6185 (0.46093)

4. Primary Outcome: Plasma Retapumulin Pharmacokinetic Parameters by Treatment at Day 5 Evaluated by Plasma Cmax After Dosing
Description: Cmax is the peak serum concentration. Low value was not calculable, and high value was 2.74 ng/mL
Time Frame: Day 5
Population: Pharmacokinetic Concentration Population - included all subjects who underwent plasma PK sampling
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days
Number analyzed (Participants) | 0 | 11
ng/mL |  | 0.5547 (0.31469)

5. Primary Outcome: Percentage of Participants With Eradication of S. Aureus Nasal Carriage at Day 12 Who Were Categorized as Persistent Carriers of S. Aureus
Description: Subjects who tested positive as persistent carriers of S. Aureus who on day 12 are negative and have been eradicated of S. Aureus.
Time Frame: Day 12
Population: Per Protocol Population: Persistent Carriers of the Intent-to-Treat (ITT) Population who Tested Positive on Screening Visit 1, 2 and 3.
Measure: Number; unit: Percentage of participants
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days | Placebo
Number analyzed (Participants) | 16 | 14 | 13
Percentage of participants | 94 | 92 | 15
Statistical Analysis 1: Comparison: Retapamulin 3 Days vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Retapamulin 5 Days vs Placebo; Test type: Superiority or Other; p < 0.001, Fisher Exact

6. Secondary Outcome: Plasma Retapumulin Pharmacokinetic Parameters, Tmax, by Treatment at Days 1 and 3
Description: Tmax - The time after administration of a drug when the maximum plasma concentration is reached, when the rate of absorption equals the rate of elimination.
Time Frame: Days 1 and 3
Population: Per Protocol Population of Intent-to-treat
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days
Number analyzed (Participants) | 16 | 10
hours
  Day 1, n=10 and 3 | 5.6000 (3.72529) | 6.9933 (5.54812)
  Day 3, n=16 and 10 | 3.8156 (2.26213) | 2.4520 (1.49694)

7. Secondary Outcome: Plasma Retapumulin Pharmacokinetic Parameters by Treatment at Day 5
Description: as for outcome 6
Time Frame: Day 5
Population: Per Protocol Population of Intent-to-treat
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days
Number analyzed (Participants) | 0 | 11
hours |  | 2.4118 (2.48003)

8. Secondary Outcome: Percentage of Participants With Eradication of S. Aureus Nasal Carriage at Days 7 and 33 Who Were Categorized as Persistent Carriers of S. Aureus
Description: Subjects who tested positive as persistent carriers of S. Aureus who on Days 7 and 33 are negative and have eradicated of S. aureus.
Time Frame: Days 7 and 33
Population: Per Protocol Population: Persistent Carriers of the Intent-to-Treat (ITT) Population who Tested Positive on Screening Visits 1, 2 and 3.
Measure: Number; unit: Percentage of participants
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days | Placebo
Number analyzed (Participants) | 16 | 14 | 13
Percentage of participants
  Day 7 | 94 | 100 | 2
  Day 33 | 75 | 86 | 4

9. Secondary Outcome: Percentage of Participants With Eradication of S. Aureus Nasal Carriage at Each Post Treatment Visit Stratified by Pharyngeal Carriage Status
Description: Comparison of nasal S. aureus eradication in persistent carrier subjects on 7, 12, and 33 days after treatment stratified by S. aureus carriage in the pharyngeal area
Time Frame: Days 1, 7, 12, and 33
Population: Per Protocol Population: Persistent Carriers of the Intent-to-Treat (ITT) Population who Tested Positive on Screening Visit 1, 2, 3, and who were Persistent Nasal carriers who were both positive and negative carriers of S. aureus in the Pharyngeal region.
Measure: Number; unit: Percentage of participants
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days | Placebo
Number analyzed (Participants) | 16 | 14 | 13
Percentage of participants
  Culture positive Day 1, Nasal eradication Day 7 | 90 | 100 | 10
  Culture negative Day 1, Nasal eradication Day 7 | 100 | 100 | 33
  Culture positive Day 1, Nasal eradication Day 12 | 90 | 86 | 10
  Culture negative Day 1, Nasal eradication Day 12 | 100 | 100 | 33
  Culture positive Day 1, Nasal eradication Day 33 | 80 | 88 | 30
  Culture negative Day 1, Nasal eradication Day 33 | 67 | 83 | 33

10. Secondary Outcome: Percentage of Participants With Nasal Recolonization With S. Aureus on Study Days 12 and 33 Who Were Persistant Carriers Who Tested Positive in the Pharyngeal Region on Days 12 and 33 But Negative in the Nasal Region on Day 7 or Days 7 and 12
Description: Percentage of subjects that were recolonized on Day 12 (D12) and Day 33 (D33) that were negative (neg.) for S. Aureus in the Pharyngeal region on days 12 or 33 and Negative in the Nasal Region on day 7 (D7) or days 7 and 12. Pharyngeal culture, PC; nasal culture, NC.
Time Frame: Days 7, 12, and 33
Population: Per Protocol Population: Persistent Carriers of the Intent-to-Treat (ITT) Population who Tested Positive on Screening Visit 1, 2, 3 and those who were NEGATIVE for Pharynegeal Carriage on Day 12 and Day 33 then recolonized.
Measure: Number; unit: Percentage of participants
Groups:
- Total: Total of all Groups
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days | Placebo | Total
Number analyzed (Participants) | 16 | 14 | 13 | 43
Percentage of participants
  PC neg. D12, NC neg. D7, Recolonized D12 | 11 | 0 | 0 | 5
  PC neg. D12, NC neg. D7 and D12, Recolonized D33 | 13 | 20 | 0 | 17
  PC neg. D33, NC neg. D7, Recolonized D12 | 0 | 0 | 100 | 6
  PC neg. D33, NC neg. D7 and D12, Recolonized D33 | 11 | 13 | 0 | 12

11. Secondary Outcome: Prevalence of S. Aureus Nasal and Pharyngeal Carriage by Visit.
Description: All participants were assessed for nasal and pharyngeal carriage at Screening Visits 1, 2, and 3. Participants were randomized into the study only if they had positive cultures at screening visit 1 and screening visit 2 and/or screening visit 3. Day 1 data were collected only for those participants who were randomized into the study.
Time Frame: Screening Visits 1 (Day -42 to Day -14), 2 (Day -11 to Day -4), and 3 (Day -11 to Day -4) and Day 1
Population: Screening Population (participants who had anterior nares swab obtained for S. aureus culture) was analyzed for Screening Visit (SV) 1. Only subjects who had positive cultures for S. aureus at SV 1 were allowed to continue to SV 2 and 3. The Safety Population (participants who received at least one dose of study drug) was analyzed at Day 1.
Measure: Number; unit: participants
Groups:
- Positive Nasal Culture for S. Aureus: Screened subjects positive for S. aureus
- Positive Pharyngeal Culture for S. Aureus: Subjects who tested positive for S. aureus in the pharyngeal region.
Arm/Group | Positive Nasal Culture for S. Aureus | Positive Pharyngeal Culture for S. Aureus
Number analyzed (Participants) | 430 | 429
participants
  Screening 1, n=430, 429 | 135 | 150
  Screening 2, n =104, 92 | 89 | 0
  Screening 3, n=92 and 58 | 74 | 0
  Day 1, n=58 and 58 | 53 | 37

12. Secondary Outcome: Number of Participants With a Nasal Culture Negative for MRSA (Methicillin-resistant S. Aureus)
Description: The number of participants who tested negative for MRSA on days 7, 12, and 33.
Time Frame: Days 7, 12, or 33.
Population: Screening Eligibility Population: only participants who provided nasal cultures at Days 7, 12, and 33 were analyzed.
Measure: Number; unit: participants
Groups:
- MRSA: Methicillin Resistant S. aureus.
Arm/Group | MRSA
Number analyzed (Participants) | 17
participants
  Day 7, n=12 | 12
  Day 12, n=14 | 13
  Day 33, n=17 | 17

13. Other Pre Specified Outcome: Percentage of Participants With Nasal Recolonization With S. Aureus on Study Days 12 and 33 Who Were Persistant Carriers Who Tested Positive in the Pharyngeal Region on Days 12 and 33 But Negative in the Nasal Region on Day 7 or Days 7 and 12
Description: All subjects were positive (pos.) for S. Aureus in the Pharyngeal region on days 12 or 33 (D12 and D33) and Negative (neg.) in the Nasal Region on day 7 (D7) or days 7 and 12. Pharyngeal culture, PC; nasal culture, NC.
Time Frame: Days 7, 12, and 33.
Population: Per Protocol Population: Persistant Carriers of the Intent-to-Treat (ITT) Population who Tested Positive on Screening Visit 1, 2, 3, and those who were Positive for Pharynegeal Carriage on Day 12 and Day 33 then recolonized.
Measure: Number; unit: Percentage of participants
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days | Placebo | Total
Number analyzed (Participants) | 16 | 14 | 13 | 43
Percentage of participants
  PC pos. D12, NC neg. D7, Recolonized D12 | 0 | 33 | 50 | 18
  PC pos. D12, NC neg. D7 and D12, Recolonized D33 | 33 | 0 | 0 | 22
  PC pos. D33, NC neg. D7, Recolonized D12 | 17 | 17 | 0 | 15
  PC pos. D33, NC neg. D7 and D12, Recolonized D33 | 40 | 25 | 0 | 30

ADVERSE EVENTS:
Arm/Group | Retapamulin 3 Days | Retapamulin 5 Days | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/19 | 0/15
Other Adverse Events (participants affected / at risk) | 6/23 | 10/19 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retapamulin 3 Days (N=23) | Retapamulin 5 Days (N=19) | Placebo (N=15)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retapamulin 3 Days (N=23) | Retapamulin 5 Days (N=19) | Placebo (N=15)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 1
Burning Sensation (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Ill-defined disorder (General disorders) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.